CLINICAL TRIAL: NCT01358422
Title: Occurrence of Bleeding and Thrombosis During Antiplatelet Therapy in Non-cardiac Surgery. A Prospective Observational Study (OBTAIN Study)
Brief Title: Occurrence of Bleeding and Thrombosis During Antiplatelet Therapy in Non-cardiac Surgery
Acronym: OBTAIN
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Collaborators: University of Leeds (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: OBTAIN
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Bleeding; Thrombosis; Cardiac Events
Keywords: Prospective observational study; major adverse cardiac events (MACE); clinically significant bleeding events; Dual anti-platelet therapy; aspirin alone therapy; non-cardiac surgery; percutaneous coronary intervention (PCI); placement of a bare metal or drug eluting stent; OBTAIN; Simon Howell; ESA; European Society of Anaesthesiology
MeSH Terms: conditions — Hemorrhage; Thrombosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- In Patients

SUMMARY:
Research questions:

1. What is the absolute risk reduction for in-hospital major adverse cardiac events (MACE) associated with the use of dual anti-platelet therapy as compared with aspirin alone in this population?
2. What is the absolute risk increase for clinically significant bleeding during the same period associated with the use of dual anti-platelet therapy as compared with aspirin alone in this population?

In brief the design of the study is as follows:

* We will study patients undergoing non-cardiac surgery within four years of coronary stenting.
* We will record the anti-platelet agents taken by patients before, during and after surgery.
* We will record cardiac and bleeding events that occur whilst the patient is in hospital.
* We will use the statistical technique of propensity scoring to match patients who have similar risk factors and who received different anti-platelet regimens.
* We will compare the incidence of cardiac events and bleeding in the matched groups.

DETAILED DESCRIPTION:
This study will compare the use of aspirin alone with dual antiplatelet therapy (i.e. aspirin and clopidogrel) in patients presenting for elective non-cardiac surgery who have undergone PCI with either bare metal stent or drug eluting stent placement in the four years prior to surgery. The absolute risk reduction in major adverse cardiac events (MACE) with dual antiplatelet therapy and the absolute risk increase for clinically significant bleeding events with dual therapy will be determined. This will allow the number needed to treat (NNT) for the prevention of MACE and the number needed to harm (NNH) for bleeding to be determined and the optimal antiplatelet therapy in this setting to be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing non-cardiac surgery within four years of percutaneous coronary intervention (PCI) with the placement of a bare metal or drug eluting stent will be included in the study.

Exclusion Criteria:

* Patients maintained on anticoagulant therapy e.g. heparin infusion before and after surgery will be excluded. (Patients receiving prophylactic doses of heparin for prevention of thromboembolic events will be eligible for inclusion.)
* Patients receiving bridging therapy with full anticoagulant does of heparin or other drugs to compensate for the withdrawal of antiplatelet drugs will be excluded.
* Patients who are anticoagulated with warfarin (INR>1.5 at the time of surgery) will be excluded.
* Patients receiving full anticoagulation with heparin for a known recent a known thromboembolic event (APPT ratio > 1.5) be excluded. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing non-cardiac surgery within four years of percutaneous coronary intervention (PCI) with the placement of a bare metal or drug eluting stent will be included in the study.
Sampling Method: Probability Sample
Enrollment: 830 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
1. MACE | In-hospital stay up to 30 days
  This study will record and analyse in-hospital adverse cardiac events. Major Adverse Cardiac Events (MACE) will be defined as a composite of:
  1. Myocardial infarction as defined by the Universal Definition of Myocardial Infarction(including cardiac arrest and cardiac death as described in this definition).
  2. PCI for a cardiac event occurring following surgery.
2. Clinically significant bleeding | In-hospital stay up to 30 days
  This study will record and analyse in-hospital clinically significant bleeding.
  Clinically Significant Bleeding Events will be defined as:
  1. Reoperation for bleeding.
  2. Gastrointestinal haemorrhage
  3. Intracranial haemorrhage
  4. Spinal/epidural haematoma. The transfusion of blood and blood products will also be recorded and compared between patients on dual antiplatelet therapy and aspirin alone.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Howell, MD, Study Chair — Sectional of Translational Anaesthetic and Surgical Sciences, University of Leeds, United Kingdom
Locations (3):
- University Hospital Carl Gustav Carus, Dresden, Germany
- Erasmus University, Rotterdam, Netherlands
- University of Leeds, Sectional of Translational Anaesthetic and Surgical Sciences, Leeds, United Kingdom

REFERENCES:
- [Background] Howell SJ, Hoeks SE, Poldermans D, West RM, Wheatcroft SB. OBTAIN: a study of the occurrence of bleeding and thrombosis during anti-platelet therapy in non-cardiac surgery. Eur J Anaesthesiol. 2011 Jun;28(6):456-9. doi: 10.1097/EJA.0b013e328344b4fc. No abstract available. PMID 21544024